CLINICAL TRIAL: NCT04393285
Title: A Phase II Study of Abemaciclib in Combination With Letrozole in Advanced, Recurrent or Metastatic Endometroid Endometrial Cancer
Brief Title: Abemaciclib and Letrozole to Treat Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-3039
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — abemaciclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abemaciclib and Letrozole (Experimental): Study treatment will consist of abemaciclib 150mg orally twice a day and letrozole 2.5mg orally once a day.
  Interventions: Drug: Abemaciclib; Drug: Letrozole

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib 150mg orally twice a day
Drug: Letrozole — Letrozole 2.5mg orally once a day

SUMMARY:
This is a phase II single arm trial to determine the percentage of patients without evidence of disease progression on abemaciclib and letrozole in advanced stage, persistent or recurrent endometrioid endometrial cancer at 6 months. Treatment will continue until either unacceptable toxicity, progression of disease, or investigator/patient request for withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have advanced (FIGO 2014 Stage III or IV), persistent, or recurrent endometrial carcinoma, which is not likely to be curable by surgery or radiotherapy. Histologic confirmation of recurrent disease is required. For cases of persistent disease, histologic confirmation of the primary disease with radiologic evidence of progression is required.
2. Patients must have endometrioid histology (all grades allowed) based on hysterectomy or biopsy specimen (Hormone receptor status is not required for enrollment).

   Sites are required to report results of previous MMR, MSI, and ER/PR status testing in Medidata Rave if available.
3. All patients must have measurable disease. Measurable disease is defined by RECIST version 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be greater than or equal to 10mm when measured by CT, MRI or caliper measurement by clinical exam; or greater than or equal to 20mm when measured by chest x-ray. Lymph nodes must be greater than or equal to 15mm in short axis when measured by CT or MRI.

   Patient must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
4. Prior chemotherapy in the adjuvant setting for Stage I, II, or III is permitted. Prior chemoradiotherapy for a pelvic recurrence is permitted.

   Note: Chemotherapy in the setting of Stage IV disease is permitted but the patient must be without evidence of disease at the completion of chemotherapy and have at least six months of progression-free survival since the completion of chemotherapy before detection of the recurrent cancer for which she is receiving treatment on this protocol.

   Prior immunotherapy and/or targeted therapy is allowed in addition to, in combination with, in lieu of, or subsequent to prior chemotherapy.

   Regardless of circumstances, no more than one prior chemotherapy regimen (including chemo-radiotherapy) is permitted, and no more than one additional systemic therapy is permitted. Hence, eligible patient may have received 0, 1, or 2 prior lines of systemic therapy and for women who received two prior lines of therapy, only one of them may have included chemotherapy.

   Patients who received prior chemotherapy, immunotherapy or targeted therapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to enrollment. A washout period of at least 21 days is required between last systemic therapy dose and initiation of therapy.

   Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and initiation of therapy.
5. Patient must be able to swallow oral medications.
6. Patient must have an ECOG performance status of 0 to 1.
7. Patients must have adequate organ and marrow function as defined below NOTE: Institutional/laboratory upper limit of normal = ULN Institutional/laboratory lower limit of normal = LLN

   Bone marrow function:
   * Absolute neutrophil count (ANC) greater than or equal to 1500/mcl
   * Platelets greater than or equal to 100,000 cells/mcl
   * Hemoglobin greater than or equal to 8 g/dL (Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after erythrocyte transfusion).

   Renal function:

   • Creatinine less than or equal to 1.5 x ULN

   Hepatic function:
   * Bilirubin less than or equal to 1.5 x ULN (Patients with Gilbert's syndrome with a total bilirubin ≤2 times ULN and direct bilirubin within normal limits are permitted).
   * ALT (alanine aminotransferase) and AST (aspartate aminotransferase) less than or equal to 3 x ULN
   * Alkaline phosphatase less than or equal to 2.5 x ULN
   * Albumin greater than or equal to 2.8 g/dL
8. Patients must have signed an approved informed consent and authorization permitting release of personal health information.
9. Patients must be at least 18 years of age.
10. Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing a highly effective form of contraception during the study treatment and for 8 weeks after stopping the treatment.

Highly effective contraception methods include combination of any of the following (NOTE: Estrogen containing contraceptives are prohibited):

* Use of oral, injected, or implanted hormonal methods of contraception or;
* Placement of an intrauterine device (IUD) or intrauterine system (IUS);
* Barrier methods of contraception: condom or occlusive cap (diaphgram or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository;
* Total abstinence or;
* Male/female sterilization. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.

Exclusion criteria

1. Patients who have previously received any CDK4/6 inhibitor.
2. Patients with clear cell, serous, carcinosarcoma, mixed histology endometrial cancers, or uterine sarcomas.
3. Known intolerance or hypersensitivity to abemaciclib or letrozole.
4. Patients who have previously received hormonal therapy for endometrial cancer.
5. Patients with concomitant invasive malignancy or a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the past five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol.
6. Patients receiving chronic treatment with systemic steroids or another immunosuppressive agent.
7. Patients with active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment, fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]). Screening is not required for enrollment.
8. Patients with a serious pre-existing medical condition(s) that would preclude participation in this study (for example: interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment (i.e. estimated creatinine clearance <30ml/min), history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or pre-existing chronic condition resulting in baseline grade 2 or higher diarrhea).
9. Patients with a known history of cardiac disease. This includes:

   * Uncontrolled hypertension, defined as systolic greater than 150mm Hg or diastolic greater than 90mm Hg despite antihypertensive medications
   * Myocardial infarction or unstable angina within 6 months prior to registration.
   * New York Heart Association (NYHA) Class II or greater congestive heart failure.
   * History of serious ventricular arrhythmia (i.e. ventricular tachycardia or ventricular fibrillation) or serious cardiac arrhythmia requiring medication, syncope of cardiovascular etiology or sudden cardiac arrest. This does not include asymptomatic atrial fibrillation with controlled ventricular rate.
   * Cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) within 6 months prior to the first date of study therapy.
10. Patients who are pregnant or breast-feeding.
11. Patients with known central nervous system metastases.
12. Patients with known human immunodeficiency virus (HIV) infection.
13. Patients with an impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of abemaciclib (i.e. ulcerative disease; uncontrolled nausea, vomiting and/or diarrhea; malabsorption syndrome; clinical signs and symptoms of gastrointestinal obstruction; and/or patients who require parenteral hydration and/or nutrition).
14. Patients who plan to receive live attenuated vaccines within 1 week of start of abemaciclib and during the study. Patients should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid vaccines.
15. Patients with active bleeding or pathologic conditions that carry high risk of bleeding such as known bleeding disorder or coagulopathy.
16. Patients with history of unprovoked venous thrombosis unless taking anticoagulation treatment for duration of trial.
17. Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 30 days prior to dosing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of protocol entry to date of first documented progression up to 6 months
  To evaluate the efficacy in terms of the probability of surviving progression free for at least 6 months (PFS at 6 mo)

SECONDARY OUTCOMES:
Response rate | From date of protocol entry to date of first response assessed up to 5 years
  To determine the proportion responding by RECIST v1.1 in patients with advanced, persistent, or recurrent endometrioid endometrial cancer
Time to disease progression or death | From date of protocol entry to date of progression or death assessed up to 5 years
  To estimate the time to disease progression or death (PFS and OS endpoints).
Toxicity Assessment of Adverse Events | Every 4 weeks assessed up to 5 years
  To describe the toxicities in patients receiving combination therapy with letrozole and abemaciclib

OTHER OUTCOMES:
Protein expression analysis of Cyclin D and E Pathway | At time of primary and secondary outcome analysis up to 5 years
  Perform multiplexed protein expression analysis at a single cell level using imaging mass cytometry (IMC), exploring the relationship to response, and assessing for longitudinal changes upon progression/relapse. Cyclin D and E Pathway: Protein expression of CCND1, CDK4, CDK6, RB1, phospho-RB1, CDKN2A, CCNE1, CCNE2, CDK2, CCND3
Protein expression analysis of Immune Cell Infiltration and activity | At time of primary and secondary outcome analysis up to 5 years
  Perform multiplexed protein expression analysis at a single cell level using imaging mass cytometry (IMC), exploring the relationship to response, and assessing for longitudinal changes upon progression/relapse. Immune cell infiltration and activity: CD45, CD3, CD8, CD4, FoxP3, PD-1, Tim-3, CTLA-4, CD25, Ki67.
Protein expression analysis of sex hormone/insulin/IGF pathway | At time of primary and secondary outcome analysis up to 5 years
  Perform multiplexed protein expression analysis at a single cell level using imaging mass cytometry (IMC), exploring the relationship to response, and assessing for longitudinal changes upon progression/relapse.
  Sex hormone/insulin/IGF pathway: Protein expression of ER (ESR1), PR, IR, IGF1R, and phospho-IGF1R/IR
Cyclin D1 3'UTR mutations | At time of primary and secondary outcome analysis up to 5 years
  Determine the frequency of Cyclin D1 3'UTR mutations and correlatioin with response.
Estradiol levels | At time of primary and secondary outcome analysis up to 5 years
  Compare the pre- and post-treatment circulating estradiol levels, and association with response.
Insulin levels | At time of primary and secondary outcome analysis up to 5 years
  Compare the pre- and post-treatment circulating insulin levels, and association with response.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Huang, MD, Study Chair — University of Virginia
Locations (29):
- United States (29):
  - University of South Alabama Mitchell Cancer Center, Mobile, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Smillow Cancer Care at Greenwich, Greenwich, Connecticut
  - Yale University, New Haven, Connecticut
  - Sylvester Comprehensive Cancer Center-Lennar Foundation Medical Center, Coral Gables, Florida
  - Sylevester Comprehensive Cancer Center-Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Center, Gainesville, Florida
  - University of Miami - Sylvester Cancer Center, Miami, Florida
  - UT Health Tower, Miami, Florida
  - Advent Health - Orlando, Orlando, Florida
  - Sylvester Comprehensive Cancer Center-Plantation, Plantation, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Lewis Cancer & Research Pavilion, Savannah, Georgia
  - University of Chicago, Chicago, Illinois
  - Baptist Healthcare System, Lexington, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Reading Hospital-McGlinn Cancer Institute, Reading, Pennsylvania
  - Abington Memorial Hospital, Willow Grove, Pennsylvania
  - Baptist Health Center Lexington, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia